CLINICAL TRIAL: NCT05201872
Title: Bacteriological Differences Between Transanal and Laparoscopic Total Mesorectal Excision for Rectal Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, Director, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: GIHSYSU-21
Record Dates: First submitted 2022-01-20; First posted 2022-01-21 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Rectum Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic surgery: Different surgical methods for rectal cancer resection
- Transanal endoscopic surgery: Different surgical methods for rectal cancer resection

SUMMARY:
The primary purpose of this study is to compare the differences of bacteriological in rectal cancer patients undergoing laparoscopic or transanal endoscopy radical resection. The secondary purpose is to compare the effects of two different surgical methods on postoperative complications.

DETAILED DESCRIPTION:
Transanal total mesorectal excision (taTME) is a new surgical procedure for total mesorectal excision (TME) by dissociating the mesorectum from the bottom through transanal endoscopic. The characteristics of TaTME are mainly summarized as transanal reverse operation, no auxiliary abdominal incision, complete mesorectal excision and specimen removal through the anus. So taTME is a natural orifice specimen extraction procedure (NOSES). Compared with traditional laparoscopy, taTME has obvious oncological and technical advantages. However, similar to NOSES, the specific surgical approach to taTME may induces bacteriological safety concerns. Whether TaTME is safe and feasible still needs strong evidence-based medical evidence. However, there have been prospective studies related to bacteriology in NOSES surgery, but there is a lack of prospective clinical studies on the issue of bacteriological diffusion during taTME surgery. Bacterial contamination of the peritoneal cavity is common in laparoscopic surgery for colorectal cancer. Although the standard NOSES procedure avoids bacteriological problems through the use of antibiotics, surgical peritoneal irrigation, and the use of sterile specimen bags, its safety remains inconclusive. Therefore, compared with conventional laparoscopic colorectal cancer surgery, taTME not only takes specimens from the natural orifice, but also requires further prospective studies on whether the incision of the intestinal wall from the mucosa during the operation will violate the aseptic principle, the aseptic safety of taTME still needs further prospective studies to confirm. Therefore, the investigators conducted a randomized controlled study to collect the abdominal and pelvic irrigation fluids in the transanal and laparoscopic TME surgery for bacteriological examination, to clarify the influence of the two different surgical methods on the intraoperative bacterial diffusion. The purpose of this study was to clarify the influence of two different surgical methods on the intraoperative bacterial spread, and to provide more evidence-based medical evidence for the safety of taTME surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary rectal carcinoma
* Single lesion
* No metastasis

Exclusion Criteria:

* History of malignant tumors
* Acute bowel obstruction, bleeding or perforation
* Tumor over 6cm in diameter or in severe adhesion with surrounded tissues
* Severe other contradictions of surgery
* Pregnant women will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 216 rectal cancer patients will be enrolled. Patients must be older than 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The positive rate of bacterial contamination of peritoneal washings | 1 years
  Bacterial contamination positive rate determined by bacterial culture of intra-operative peritoneal washings

SECONDARY OUTCOMES:
Postoperative complications | a month
  Determine whether patients have postoperative complications after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China